CLINICAL TRIAL: NCT00003898
Title: The Use of Supplemental Oral Glutamine (GLN) to Decrease Morbidity in Patients Undergoing Stem Cell Transplantation: A Pediatric Blood and Marrow Transplant Consortium Study
Brief Title: Glutamine in Treating Side Effects in Children Who Are Undergoing Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Barbara Bambech, MD, Roswell Park Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000067069; RPCI-RP-9810
Record Dates: First submitted 1999-11-01; First posted 2004-06-17 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Oral Complications; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: unspecified childhood solid tumor, protocol specific; oral complications
MeSH Terms: interventions — Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: glutamine — Oral

SUMMARY:
RATIONALE: Glutamine may be able to decrease inflammation of the mouth and digestive system in children who are undergoing stem cell transplantation.

PURPOSE: Randomized double-blinded phase II trial to study the effectiveness of glutamine in reducing inflammation of the mouth and digestive system in children who are undergoing peripheral stem cell transplantation.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of supplemental oral glutamine in reducing the severity and duration of mucositis in children undergoing stem cell transplantation. II. Determine the safety of this regimen in these patients. III. Determine serum glutamine levels achieved during this regimen in these patients.

OUTLINE: This is a randomized, double blind, multicenter study. Patients are stratified according to inclusion of total body irradiation in the conditioning regimen (yes vs no). Patients receive either oral glutamine or oral placebo (glycine) twice a day beginning on the day of admission for the stem cell transplant and continuing for 28 days or until hospital discharge, whichever is first.

PROJECTED ACCRUAL: A total of 120 patients (60 per arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Undergoing allogeneic or autologous stem cell transplant (including bone marrow, cord blood, or peripheral blood stem cells) Conditioning regimen must have at least 50% risk of grade III or IV mucositis No grade III or IV hepatic toxicity

PATIENT CHARACTERISTICS: Age: 1 to 21 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: See Disease Characteristics Renal: Not specified Other: No grade III or IV toxicity at admission for stem cell transplant No altered mental status

PRIOR CONCURRENT THERAPY: No concurrent vancomycin paste or nonabsorbable antibiotics

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 1999-01; Primary Completion 2003-06 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Jean Bambach, MD, Study Chair — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Simmons Cancer Center - Dallas, Dallas, Texas

REFERENCES:
- [Result] Aquino VM, Harvey A, Garvin J, et al.: The use of supplemental glutamine to decrease morbidity in children undergoing stem cell transplantation: a Pediatric Blood and Marrow Transplant Consortium study. [Abstract] 2004 Pediatric Academic Societies' Annual Meeting, May 1-4, San Francisco, California. A-1627, 2004. Availabel online Last accessed August 29, 2005.
- [Result] Aquino VM, Harvey AR, Garvin JH, Godder KT, Nieder ML, Adams RH, Jackson GB, Sandler ES. A double-blind randomized placebo-controlled study of oral glutamine in the prevention of mucositis in children undergoing hematopoietic stem cell transplantation: a pediatric blood and marrow transplant consortium study. Bone Marrow Transplant. 2005 Oct;36(7):611-6. doi: 10.1038/sj.bmt.1705084. PMID 16086046